CLINICAL TRIAL: NCT06997718
Title: Evaluation of the Effects of the Product RV5075A-MF6793 in Diabetic Patients Presenting Foot Xerosis and Superficial Fissures, an Exploratory Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RV5075A20240673
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Xerosis

STUDY DESIGN:
Intervention Model Description: The subjects are randomly divided in two groups, according to the randomization list, where one group applies the test product (product code: RV5075A), and another group applies comparative product (product code: CO5075A).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: RV5075A MF6793
- Comparative group (Active Comparator)
  Interventions: Other: CO5075A

INTERVENTIONS:
Other: RV5075A MF6793 — Twice daily applications on both feet. The product will be applied according to randomization on the entire feet in a sufficient amount.
  Arms: Test group
Other: CO5075A — Twice daily applications on both feet. The product will be applied according to randomization on the entire feet in a sufficient amount.
  Arms: Comparative group

SUMMARY:
This exploratory study is meant to assess the efficacy of a product in diabetic patients presenting foot xerosis and superficial fissures This exploratory study will be conducted as randomized, comparative study in parallel groups. In order to perform this clinical study, 60 female/male subjects, aged between 18 and 75 years old, with controlled type 1 or 2 diabetes and presenting foot xerosis and superficial fissures, are enrolled.

The subjects are randomly divided in two groups, (Group I or Group II), where one group applies the test product and another group applies comparative product.

The subjects apply the investigational/comparator products to both feet, twice a day, in the mornings and evenings, for 28 consecutive days.

3 visits are planned :

* Visit 1: Inclusion (D1)
* Visit 2: Intermediate visit (D5 ±2)
* Visit 3: End-of-study visit (D28 ±2)

ELIGIBILITY:
Main Inclusion criteria:

* Gender: Male/Female;
* Age: 18 to 75 years old;
* Presenting skin phototype between I and IV according to the Fitzpatrick phototyping scale;
* Presenting controlled type 1 or 2 diabetes;
* Presenting xerosis intensity on feet is rated as 6 according to the Xerosis Assessment Scale (XAS).

Main Non-inclusion criteria:

* Subject with uncontrolled diabetes and/or with diabetes complications
* Subjects with any foot condition or medical history liable to interfere with the evaluation of the efficacy or cutaneous tolerance of the investigational products according to the investigator's assessment
* Topical or oral treatment established or modified during the previous weeks or planned to be established or modified during the study, liable to interfere with the evaluation of the efficacy or cutaneous tolerance of the investigational products according to the investigator's assessment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Xerosis intensity on both feet with XAS (Xerosis Assessment Scale) | Before (Day 1 Visit 1), and after 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application
  Evaluation performed by the investigator, giving 1 XAS score for both feet/patient (9 points scale, from 0 = Normal skin, to 8 =Skin with deep fissures).
Evolution of superficial fissures intensity on both feet with VAS (Visual Analog Scale) | After 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application compared to baseline (Day 1, Visit 1)
  Evaluation performed by the investigator, giving 1 VAS score for both feet/patient (continuous sliding scale from 0 mm = no repair/no improvement to 100 mm = complete repair/full improvement).
Evolution of superficial fissures intensity on a target fissure with VAS (Visual Analog Scale) | After 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application compared to baseline (Day 1, Visit 1)
  Evaluation performed by the investigator specifically on the target fissure identified at the inclusion visit, on VAS (continuous sliding scale from 0 mm = no repair/no improvement to 100 mm = complete repair/full improvement).
Quality of Life evaluation by the patient | Before (Day 1, Visit 1), and after 28 (Visit 3) consecutive days of products' application
  Filling by the patient of a 13-questions questionnaire about their quality of life related to their feet condition.
Global soothing effect evaluation on feet | After the first application (Day 1, Visit 1), and after 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application
  The global soothing is assessed by each subject using a VAS (continuous sliding scale from 0 mm = no relief/no soothing effect to 100 mm = complete relief/total soothing effect)
Intensity of pruritus/itchiness on feet | Before (Day 1, Visit 1) and immediately after the first application (Day 1, Visit 1), and after 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application
  The evolution of pruritus intensity on feet is assessed by each subject using a VAS (continuous sliding scale from 0 mm = no itching or pruritus at all, to 100 mm = extreme itching, unbearable)
Intensity of tingling on feet | Before (Day 1, Visit 1) and immediately after the first application (Day 1, Visit 1), and after 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application
  The evolution of tingling intensity on feet is assessed by each subject using a VAS (continuous sliding scale from 0 mm = no tingling sensation, to 100 mm = intense tingling, very uncomfortable)
Intensity of tightness on feet | Before (Day 1, Visit 1) and immediately after the first application (Day 1, Visit 1), and after 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application
  The evolution of tightness intensity on feet is assessed by each subject using a VAS (continuous sliding scale from 0 mm = no tightness at all, to 100 mm = extreme tightness, uncomfortable)
Intensity of pain on feet | Before (Day 1, Visit 1) and immediately after the first application (Day 1, Visit 1), and after 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application
  The evolution of pain intensity on feet is assessed by each subject using a VAS (continuous sliding scale from 0 mm = no pain at all, to 100 mm = extreme pain, debilitating)
Skin hydration | Before (Day 1, Visit 1) and after 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application
  Skin capacitance is assessed instrumentally by an expert, on the selected foot of each subject
Standardized photographs of the target fissure of each subject to visually assess the evolution of the target fissure. | Before (Day 1, Visit 1) and after 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application
Cosmetic satisfaction and perceived effect evaluation questionnaire | After the first application (Day 1, Visit 1), and after 5 (Visit 2), 15 (at home) and 28 (Visit 3) consecutive days of products' application
  Filling by the patient of a subjective evaluation questionnaire considering their cosmetic acceptability, and perceived efficacy towards the investigational/comparator product
Standardized photograph of the selected foot of each subject is taken for illustrative purposes | Before (Day 1, Visit 1) and after 5 (Visit 2) and 28 (Visit 3) consecutive days of products' application
Compliance of the subject to the product | During the entire course of the study, from inclusion visit (Day 1), to the end-of-study visit (Day 28).
  Subjects fill in a subject diary (daily log) during the course of the study to record their compliance to the product.
Global assessment of the tolerance | At the end of the study (after 28 consecutive days of products' twice-daily application), or premature withdrawal
  Global assessment of the tolerance is assessed by the investigator for each subject at the end of the study considering all individual adverse events and their characteristics, based on a 5-point scale (from excellent tolerance to bad tolerance).

CONTACTS AND LOCATIONS:
Locations (1):
- Inovapotek, Porto, Portugal